CLINICAL TRIAL: NCT00434798
Title: Campylobacter Jejuni Challenge Model Development: Dose Ranging Study
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: University of Vermont (Other)
Collaborators: Naval Medical Research Center (U.S. Federal Agency); TD Vaccines A/S (Industry)
Responsible Party: Beth Kirkpatrick, M.D., Principal Investigator, University of Vermont
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: NMRC.2006.0009
Record Dates: First submitted 2007-02-06; First posted 2007-02-13 (Estimated); Last update posted 2008-06-05 (Estimated); Status verified 2008-06

CONDITIONS: Campylobacter Infections
Keywords: Campylobacter infections
MeSH Terms: conditions — Campylobacter Infections

INTERVENTIONS:
Biological: Campylobacter jejuni strains CG8421 and BH-01-0142 — Campylobacter jejuni strains CG8421 and BH-01-0142 at a single dose. Dosing will be based on attack rate, to achieve a 75% attack rate. Anticipate use of 10^6-10^9 CFU

SUMMARY:
The primary objective of this study is to establish a human Campylobacter jejuni infection model with the following characteristics:

1. Safe application

   1. Infectious period risk mitigated by close monitoring and prospectively applied early treatment criteria
   2. Potential post-infectious sequelae risk mitigated by appropriate strain and host selection
2. Campylobacteriosis attack rate of at least 75%

Secondary objectives are to determine humoral, cell-mediated, and mucosal immune responses in the newly established human C. jejuni infection model and evaluate short-term (< 3 mo) protection upon repeat exposure to homologous C. jejuni strain and assess immune responses associated with protection.

ELIGIBILITY:
Inclusion Criteria:

* Male or female between 18 and 50 years of age, inclusive.
* General good health, without significant medical illness, abnormal physical examination findings or clinical laboratory abnormalities as determined by principal investigator or principal investigator in consultation with the medical monitor and sponsor.
* Demonstrate comprehension of the protocol procedures and knowledge of Campylobacter illness by passing a written examination (pass grade ≥ 70%)
* Willing to participate after informed consent obtained.
* Available for all planned follow-up visits.
* Negative urine pregnancy test at screening and a negative urine pregnancy test on the day of admittance to the inpatient phase for all female subjects.

Exclusion Criteria:

* Presence of a significant medical condition, (e.g. psychiatric conditions or gastrointestinal disease, such as peptic ulcer, symptoms or evidence of active gastritis, inflammatory bowel disease, irritable bowel syndrome, alcohol or illicit drug abuse/dependency), or other laboratory abnormalities which in the opinion of the investigator precludes participation in the study.
* Immunosuppressive illness, IgA deficiency (below the normal limits), or antihistamine use within 48 h of admission or during inpatient period.
* Positive serology results for HIV, HBsAg, or HCV antibodies.
* Significant abnormalities in screening lab hematology, serum chemistry, as determined by PI or PI in consultation with the medical monitor and sponsor.
* Use of any medication known to affect the immune function (e.g., corticosteroids and others) within 30 days preceding receipt of the challenge inoculum or planned use during the active study period.
* Are not capable of fully informed consent (e.g. cannot read or write English)
* Personal or documented family history of an inflammatory arthritis such as reactive arthritis, Reiter's syndrome, ankylosing spondylitis, rheumatoid arthritis, or Guillain-Barré syndrome (would not include osteoarthritis or vague history of arthritis relatively late in adulthood).
* Evidence of neurologic abnormalities (specifically extremity weakness, abnormal deep tendon reflexes, symmetric sensory abnormalities - vibratory, light touch, and proprioception).
* Evidence of inflammatory arthritis on exam and/or HLA-B27 positive.
* Allergy or prior intolerance to either azithromycin or fluoroquinolones.
* Fewer than 3 stools per week or more than 3 stools per day as the usual frequency, loose or liquid stools other than on an occasional basis.
* Regular use of laxatives or any agent that increase gastric pH (regular defined as at least weekly).
* A recent fever in the 2 weeks prior to time of challenge.
* Use of antibiotics during the 7 days before bacterial dosing or proton pump inhibitors, H2 blockers, or antacids within 48 hours of dosing.
* Use of any investigational product within 30 days preceding the receipt of the challenge inoculum, or planned use during the active study period.
* History of diarrhea in the 2 weeks prior to planned inpatient phase
* Stool culture (collected no more than 1 week prior to admission) positive for Campylobacter, other bacterial enteric pathogens (Salmonella, Shigella, or enterohemorrhagic E. coli), or intestinal parasites.
* Have household contacts who are <2 years old or >80 years old or infirmed or immunocompromised (for reasons including corticosteroid therapy, HIV infection, cancer chemotherapy, or other chronic debilitating disease).
* Work as either a health care personnel with direct patient care, daycare center (for children or the elderly) personnel, or food handlers. Food handlers include individuals who work in restaurants, cafeterias, and retail stores/supermarkets that feature produce, salad bars, and/or deli sections.
* History of microbiologically confirmed Campylobacter infection
* Immunologic evidence of Campylobacter exposure:

  * serologic evidence of prior Campylobacter infection [defined as homologous strain Campylobacter-specific anti-glycine extract (GE) IgA OD650 > 0.5 at > 1:1,000 dilution]
  * cell mediated immune response evidence of prior Campylobacter infection [in vitro stimulation of PBMC with WC antigen (formalin-fixed homologous strain Campylobacter whole cells) with supernatant IFN-Gamma ≥ 500pg/ml]
* Travel to countries with high Campylobacter rates (to include Asia, Africa, and Central and South America) within two years prior to dosing.
* History of vaccination for or ingestion of Campylobacter.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 50 (Estimated)
Dates: Start 2007-02; Primary Completion 2008-10 (Estimated); Study Completion 2008-10 (Estimated)

PRIMARY OUTCOMES:
Establish a safe challenge model of Campylobacter jejuni | October 2008

SECONDARY OUTCOMES:
Measurement of the human immune response to Campylobacter jejuni infection | October 2008

CONTACTS AND LOCATIONS:
Locations (1):
- University of Vermont College of Medicine, Burlington, Vermont, United States